CLINICAL TRIAL: NCT03540160
Title: An Open-Label Long-Term Safety Study of Serlopitant for the Treatment of Pruritus
Brief Title: Study of the Long Term Safety of Serlopitant for the Treatment of Pruritus (Itch)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No longer pursuing development of serlopitant
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTI-107; 2017-004211-40 (EudraCT Number)
Record Dates: First submitted 2018-04-05; First posted 2018-05-30 (Actual); Results first posted 2020-11-30 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pruritus; Prurigo Nodularis; Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic; Psoriasis | interventions — serlopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: 5 mg Serlopitant Tablets (Experimental): Serlopitant Tablets
  Interventions: Drug: 5 mg Serlopitant Tablets

INTERVENTIONS:
Drug: 5 mg Serlopitant Tablets — Serlopitant Tablets
  Other Names: VPD-737

SUMMARY:
Study of the long term safety of serlopitant for the treatment of pruritus in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older at consent.
* Pruritus associated with prurigo nodularis, atopic dermatitis, or psoriasis.
* Female subjects of childbearing potential must be willing to practice highly effective contraception until 5 weeks after last dose of study drug.
* Willing and able to comply with study visits and study related requirements including providing written informed consent.

Exclusion Criteria:

* Malignancy within 5 years prior to enrollment (exception for non-melanoma cutaneous malignancies).
* Any known major psychiatric diagnosis, such as major depressive disorder, bipolar disorder, schizophrenia, psychotic disorder, intellectual disability, severe alcohol use disorder, which may confound the assessment of serlopitant safety or efficacy, or interfere with the subject's ability to comply with protocol-mandated activities, within 3 years prior to enrollment.
* Untreated or inadequately treated thyroid, adrenal, or pituitary nodules or disease, or history of thyroid malignancy; or the prescense of any medical condition or disability, that could interfere with the assessment of safety in this study or compromise the safety of the subject.
* Investigational therapy within 4 weeks or 5-half-lives prior to enrollment (whichever is longer) or expected participation in another clinical study involving an investigational product or device during the subject's participation in this study.
* Treatment with other neurokinin-1 receptor (NK1-R) antagonists (e.g., aprepitant, fosaprepitant, rolapitant) within 4 weeks.
* Treatment with strong cytochrome P450 3A4 inhibitors within 4 weeks.
* Currently pregnant or breastfeeding or planning to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (85):
- United States (46):
  - Study Site 504, Birmingham, Alabama
  - Study Site 204, Fremont, California
  - Study Site 383, North Hollywood, California
  - Study Site 356, San Diego, California
  - Study Site 514, Santa Ana, California
  - Study Site 501, Aventura, Florida
  - Study Site 210, Coral Gables, Florida
  - Study Site 534, Fort Lauderdale, Florida
  - Study Site 531, Miami, Florida
  - Study Site 222, North Miami Beach, Florida
  - Study Site 510, Newnan, Georgia
  - Study Site 388, Skokie, Illinois
  - Study Site 228, Louisville, Kentucky
  - Study Site 527, New Orleans, Louisiana
  - Study Site 525, Glenn Dale, Maryland
  - Study Site 506, Ann Arbor, Michigan
  - Study Site 515, Detroit, Michigan
  - Study Site 371, Saint Joseph, Missouri
  - Study Site 528, St Louis, Missouri
  - Study Site 227, Omaha, Nebraska
  - Study Site 526, Henderson, Nevada
  - Study Site 201, East Windsor, New Jersey
  - Study Site 529, Verona, New Jersey
  - Study Site 507, Brooklyn, New York
  - Study Site 508, Buffalo, New York
  - Study Site 500, New York, New York
  - Study Site 517, New York, New York
  - Study Site 341, High Point, North Carolina
  - Study Site 516, Bexley, Ohio
  - Study Site 509, Cleveland, Ohio
  - Study Site 524, Dublin, Ohio
  - Study Site 112, Tulsa, Oklahoma
  - Study Site 523, Philadelphia, Pennsylvania
  - Study Site 522, Pittsburgh, Pennsylvania
  - Study Site 345, Johnston, Rhode Island
  - Study Site 343, Spartanburg, South Carolina
  - Study Site 511, Knoxville, Tennessee
  - Study Site 365, Austin, Texas
  - Study Site 520, Bellaire, Texas
  - Study Site 502, Dallas, Texas
  - Study Site 224, Houston, Texas
  - Study Site 359, Pflugerville, Texas
  - Study Site 226, Webster, Texas
  - Study Site 336, Richmond, Virginia
  - Study Site 806, Spokane, Washington
  - Study Site 532, Morgantown, West Virginia
- Austria (3):
  - Study Site 649, Graz
  - Study Site 648, Linz
  - Study Site 650, Vienna
- Germany (19):
  - Study Site 623, Bad Bentheim
  - Study Site 607, Berlin
  - Study Site 641, Berlin
  - Study Site 600, Bielefeld
  - Study Site 617, Bochum
  - Study Site 608, Bonn
  - Study Site 642, Buxtehude
  - Study Site 606, Dresden
  - Study Site 621, Erlangen
  - Study Site 602, Frankfurt am Main
  - Study Site 639, Hamburg
  - Study Site 605, Heidelberg
  - Study Site 611, Leipzig
  - Study Site 620, Mahlow
  - Study Site 614, Mainz
  - Study Site 601, Münster
  - Study Site 618, Osnabrück
  - Study Site 615, Selters
  - Study Site 643, Stuttgart
- Poland (17):
  - Study Site 636, Bydgoszcz
  - Study Site 628, Iwonicz-Zdrój
  - Study Site 633, Krakow
  - Study Site 624, Krakow
  - Study Site 635, Krakow
  - Study Site 629, Lodz
  - Study Site 631, Olsztyn
  - Study Site 625, Osielsko
  - Study Site 645, Poznan
  - Study Site 644, Poznan
  - Study Site 634, Rzeszów
  - Study Site 638, Szczecin
  - Study Site 632, Torun
  - Study Site 627, Warsaw
  - Study Site 637, Wroclaw
  - Study Site 630, Wroclaw
  - Study Site 647, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 120 sites from 15 March 2018 to 08 April 2020. All participants who met the study entry criteria received daily oral doses of serlopitant 5 mg tablet.
Pre-assignment Details: Subjects attended a screening visit before receiving their first dose. All subjects underwent inclusion exclusion criteria assessment and all eligible subjects signed the informed consent before undergoing any study-related procedures.
Groups:
- Serlopitant 5 mg: Subjects received serlopitant 5 mg tablet once daily orally from Baseline Visit (Study Day 1) until the Week 52 Visit.
Period: Overall Study
Arm/Group | Serlopitant 5 mg
Started | 558
Completed | 179
Not Completed | 379
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 8
Not completed — Lack of Efficacy | 60
Not completed — Pregnancy | 1
Not completed — Adverse Event | 20
Not completed — Withdrawal by Subject | 68
Not completed — COVID-19 | 2
Not completed — Study Closure | 10
Not completed — Lost to Follow-up | 18
Not completed — Sponsor decision | 191

BASELINE CHARACTERISTICS:
Population: Nine subjects were excluded from the safety population (all from US) due to no evidence of subject dosing and/or no post-Baseline assessment/treatment emergent adverse event.
Arm/Group | Serlopitant 5 mg
Number analyzed (Participants) | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 351
  Male | 198
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 80
  White | 442
  More than one race | 7
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Treatments emergent adverse events (TEAEs) and serious adverse events (SAEs) were recorded from the first study drug administration through the follow-up visit. Severity of all AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03. During the period between informed consent and first study drug dose, only SAEs caused by a protocol-mandated intervention were collected.
Time Frame: From baseline until the Follow-up (F/U) visit which occurred 35 days (+ 7 days) after the Week 52 visit or the last dose of study drug for subjects who discontinued study drug early.
Population: Safety population: included all treated participants with at least one postbaseline assessment or a reported TEAE.
  No statistical analyses were performed for this end point
Measure: Count of Participants; unit: Participants
Arm/Group | Serlopitant 5 mg
Number analyzed (Participants) | 549
Participants
  Subjects with any TEAE | 325
  Subjects with any related TEAE | 55
  Subjects with any SAE | 45
  Subjects with any related SAE | 1
  Subjects who died | 0
  Subjects who discontinued study drug due to TEAE | 28

ADVERSE EVENTS:
Time Frame: From baseline until the F/U visit which occurred 35 days (+ 7 days) after the Week 52 visit or the last dose of study drug for subjects who discontinued study drug early
Description: Subjects received serlopitant 5 mg tablet once daily orally.
Arm/Group | Serlopitant 5 mg
All-Cause Mortality (participants affected / at risk) | 0/549
Serious Adverse Events (participants affected / at risk) | 45/549
Other Adverse Events (participants affected / at risk) | 36/549
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serlopitant 5 mg (N=549)
Arterial occlusive disease (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Hernia hiatus repair (Surgical and medical procedures) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Adjustment disorder with anxiety (Psychiatric disorders) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Craniofacial fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Anticoagulation drug level below (Investigations) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Ventricular asystole (Cardiac disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Neurodegenerative disorder (Nervous system disorders) | 3
Radiculopathy (Nervous system disorders) | 1
Corneal perforation (Eye disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Pancreatic disorder (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Abscess jaw (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Diarrhoea infectious (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serlopitant 5 mg (N=549)
Nasopharyngitis (Infections and infestations) | 36

LIMITATIONS AND CAVEATS:
Due to a corporate decision to no longer pursue an indication of treatment for pruritus, and further to terminate the development program for serlopitant, the study was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT03540160/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT03540160/SAP_001.pdf